CLINICAL TRIAL: NCT00427661
Title: A Pilot Study of Allogeneic Hematopoietic Stem Cell Transplantation for Patients With High Risk Hemoglobinopathy Using a Non-Myeloablative Preparative Regimen to Achieve Stable Mixed Chimerism
Brief Title: A Pilot Study of HSCT for Patients With High-risk Hemoglobinopathy Using a Nonmyeloablative Preparative Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, MD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #0504048
Record Dates: First submitted 2007-01-18; First posted 2007-01-29 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Sickle Cell Disease; Thalassemia; Hemoglobinopathies
Keywords: Sickle Cell Disease; Thalassemia; Hemoglobinopathies
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Hemoglobinopathies | interventions — Busulfan; fludarabine; Cyclosporine; fludarabine phosphate; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AHCT in High Risk SCD (Other): Intervention: Busulfan; Fludarabine; cyclosporine A and MMF
  Interventions: Other: Busulfan; Fludarabine; cyclosporine A and MMF

INTERVENTIONS:
Other: Busulfan; Fludarabine; cyclosporine A and MMF — Hematopoietic stem cell transplantation from a matched sibling or unrelated donor following a reduced intensity conditioning regimen
  Other Names: Busulfex, Fludara, Gengraf, CellCept

SUMMARY:
Hypothesis 1: A novel nonmyeloablative condition regimen will be safe and efficacious in producing stable donor chimerism and cure of severe hemoglobinopathy.

Hypothesis 2: Stable donor chimerism will result in amelioration of cerebral vasculopathy, improved cerebral perfusion and neurocognitive function.

Specific Aim 1: Study the safety and efficacy of a novel non-toxic conditioning regimen for HSCT for patients with severe hemoglobinopathies and the kinetics of lineage specific chimerism after HSCT

We will test our hypothesis that a novel nonmyeloablative condition regimen will be safe and efficacious in producing stable donor chimerism and cure of severe hemoglobinopathy:

Specific Aim 2: Optimize the immunosuppressive regimen for HSCT patients through a thorough understanding of the pharmacokinetics of Busulfan (BU) and mycophenolate mofetil (MMF) in the patient population. This will involve:

1. Determine the pharmacokinetics of intravenously and orally administered MMF and intravenous BU in patients receiving HSCT.
2. Determine the relationship of Area under the curve (AUC) of BU and mean trough concentrations of mycophenolic acid (MPA) to engraftment and graft versus host disease (GVHD).
3. Determine the relationship of Area under the curve (AUC) and steady state concentration of BU to engraftment at day 30 and 1 year post HSCT.

Specific Aim 3: Study the effect of complete or partial donor chimerism on silent and overt cerebral vasculopathy, and neurocognitive functioning in patients with SCD undergoing HSCT. We will test our hypothesis that stable donor chimerism will result in improvement in cerebral vasculopathy and neurocognitive function. This will include.

1. Determine effect of transplantation silent and overt cerebral vasculopathy by comparison MRA and TCD 1 year after HSCT to pre-HSCT studies.
2. Determine effect on HSCT on neurocognitive function. Specific Aim 4: To determine the rate of T cell immune reconstitution in children with sickle cell disease following myeloablative compared to nonmyeloablative stem cell transplantation, using immunophenotyping assays, CDR3 spectratyping TREC analysis, and measurement of T cell specific donor engraftment.

DETAILED DESCRIPTION:
Severe hemoglobinopathies such as sickle cell disease (SCD) and Thalassemia are associated with considerable morbidity, organ damage and premature mortality. Allogeneic hematopoietic stem cell transplantation (HSCT) is the only therapy that can cure a hemoglobinopathy. The applicability of HSCT for hemoglobinopathies is limited by the paucity of suitable donors, and risk of early regimen-related toxicity and the late effects. Reduction of the dose of myelotoxic drugs in preparative regimens prior to HSCT has the potential to increase the applicability of this curative option for patients with hemoglobinopathies. We hypothesize that a preparative regimen that maximizes host immunosuppression without myeloablation will be well tolerated and sufficient for engraftment of donor hematopoietic stem cells in patients with severe hemoglobinopathies. The long term objective of this research is to develop novel, less toxic approaches to HSCT for patients with severe hemoglobinopathies. Specific aims: 1. To evaluate the safety and efficacy of a novel nontoxic nonmyeloablative approach to hematopoietic stem cell transplantation for hemoglobinopathies. 2. To optimize the immunosuppressive regimen for HSCT patients through a thorough understanding of the pharmacokinetics of Busulfan (BU) and Mycophenolic acid (MPA) 3. To determine the effect of partial or complete donor chimerism on cerebral vasculopathy in patients with SCD. 4. To determine the rate of T cell immune reconstitution in children with sickle cell disease following myeloablative compared to nonmyeloablative stem cell transplantation, using immunophenotyping assays, CDR3 spectratyping TREC analysis, and measurement of T cell specific donor engraftment. Subjects meeting eligibility criteria in whom an human leukocyte antigen matched, partially mismatched related or unrelated donor of bone marrow or umbilical cord blood will receive a HSCT after a nonmyeloablative preparative regimen consisting of BU, Fludarabine (FLU), total lymphoid radiation and Anti-Thymocyte globulin followed by prophylaxis against graft versus host disease with cyclosporine A and MMF. Patients will be studied for survival, cure of hemoglobinopathy, absence of severe regimen related toxicity and graft versus host disease. The relationship of engraftment, survival and Graft versus host disease to kinetics of lineage specific donor chimerism and area under the curve for Mycophenolic acid and Busulfan will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SCD 0-35 years of age with an HLA-identical or 1 HLA antigen mismatched bone marrow or up to 2 HLA antigen mismatched umbilical cord blood (UCB) donor with one or more of the following:

  * Stroke, CNS hemorrhage or a neurologic event lasting longer than 24 hours, or abnormal cerebral MRI or cerebral arteriogram or MRI angiographic study and impaired neuropsychological testing,
  * Acute chest syndrome with a history of recurrent hospitalizations or exchange transfusions,
  * Recurrent vaso-occlusive pain 3 or more episodes per year for 3 years or more years or recurrent priapism,
  * Impaired neuropsychological function and abnormal cerebral MRI scan,
  * Stage I or II sickle lung disease,
  * Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate [GFR] 30-50% of the predicted normal value),
  * Bilateral proliferative retinopathy and major visual impairment in at least one eye,
  * Osteonecrosis of multiple joints with documented destructive changes,
  * Requirement for chronic transfusions but with RBC alloimmunization >2 antibodies during long term transfusion therapy.
  * Patients with transfusion dependent Thalassemia 0-35 years of age with an HLA-identical or 1 HLA antigen mismatched bone marrow or up to 2 HLA antigen mismatched UCB donor.
* Second Transplants

  * Patients with sickle cell disease or Thalassemia who have failed to engraft or have autologous recovery are eligible for this protocol.
  * Patients must meet above criteria.
  * If first transplant was a non-myeloablative regimen, the second transplant can occur at any time.
  * If the first transplant was a myeloablative regimen, then the second transplant must be > 6 months from the first transplant.

Exclusion Criteria:

* Patients with one or more of the following:

  * Karnofsky or Lansky performance score <70,
  * Acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on biopsy,
  * Stage III-IV lung disease,
  * GFR<30% predicted normal values.
  * Pregnant or lactating females.
* Active serious infection whereby patient has been on intravenous antibiotics for one week prior to study entry. Any patient with AIDS or ARC or HIV seropositivity. Any patient with invasive aspergillums infection within one year of study entry.
* Psychologically incapable of undergoing BMT with associated strict isolation or documented history of medical non-compliance.
* Patients not able to receive TLI due to prior radiation therapy.

Donor Inclusion Criteria

* Donor must be in good health based on review of systems and results of physical examination.
* Donor must have a normal hemoglobin, white count, platelet count and PTT.
* Female donors of childbearing potential must have a negative pregnancy test.

Donor Exclusion Criteria

* Donor has active infection (including HIV, hepatitis).
* Donor is a lactating female.

Donor Selection

In the case where more than one donor meets the eligibility criteria, donor selection will be guided by the following considerations:

* HLA A, B, DRB1 identical sibling donor is preferable to an unrelated donor
* Homozygous normal donor is preferable to heterozygote (carrier)
* ABO-compatible donor is preferable to ABO-incompatible donor
* Younger donor is preferable to older
* Cytomegalovirus seronegative donor is preferable to CMV seropositive donor, if the patient is CMV negative

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2002-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AHSC in Severe SCD: The patient population for this study included severe SCD patients, both pediatric and adult, who did not have end-organ failure, and met all of the eligibility criteria.
Period: Overall Study
Arm/Group | AHSC in Severe SCD
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AHSC in Severe SCD
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Development of GVHD Within 1 Year of BMT
Description: GVHD is assessed by physical exam, bloodwork and biopsy.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | AHSC in Severe SCD
Number analyzed (Participants) | 7
participants | 2

2. Primary Outcome: Engraftment at 1 Year Post BMT.
Description: Measurement of total PBMC chimerism
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | AHSC in Severe SCD
Number analyzed (Participants) | 7
participants | 6

3. Secondary Outcome: Incidence of Grade 2-4 Acute GVHD.
Time Frame: 100 days
Measure: Number; unit: participants with grade 2-4 AGVHD
Groups:
- Experimental: Busulfan, Fludarabine, Cyclosporine, MMF
Arm/Group | Experimental
Number analyzed (Participants) | 8
participants with grade 2-4 AGVHD | 1

ADVERSE EVENTS:
Arm/Group | AHSC in Severe SCD
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AHSC in Severe SCD (N=8)
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 — 21 year old female patient developed complications related to sickle cell disease associated progressive pulmonary arterial hypertension and died 10 months post BMT.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AHSC in Severe SCD (N=8)
Seizure (Nervous system disorders) | 1/7 (1) — Seizure day+11 secondary to low level of phenytoin (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270.)
Headache (Nervous system disorders) | 1 (1) — headache day +1-+4, post transplant, requiring analgesics (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270)
Line related bacteremia (Infections and infestations) | 1 (1) — line related bacteremia with Rhizobium radiobactor d100 (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270.
Pancreatitis (Gastrointestinal disorders) | 1 (1) — Mild pancreatitis Day +109 (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270)
Infection (Infections and infestations) | 1 (1) — Dermatomal herpes zoster Parainfluenza A infection (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270)
Line related bacteremia (Infections and infestations) | 1 (1) — Line related bacteremia d244 (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270)
Poor oral intake (Gastrointestinal disorders) | 2 (2) — Required transient parenteral alimentation (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) — Hemoglobinuria immediately following stem cell transplant the resolved within 48 hours (Krishnamurti et al., 2008. Biol Blood Marrow Transplant 14:1270)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No